CLINICAL TRIAL: NCT04513197
Title: NEW ONSET ENDOCRINE DYSFUNCTION AFTER ACUTE PANCREATITIS(PANCREATICOGENIC DIABETES MILLETUS - TYPE 3C)
Brief Title: NEW ONSET ENDOCRINE DYSFUNCTION AFTER ACUTE PANCREATITIS
Acronym: APPDM
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Asian Institute of Gastroenterology, India (Other)
Responsible Party: Principal Investigator, Mohan Ramchandani, Dr, Asian Institute of Gastroenterology, India
Other Study IDs: NODAP
Record Dates: First submitted 2020-08-11; First posted 2020-08-14 (Actual); Last update posted 2020-08-14 (Actual); Status verified 2020-08

CONDITIONS: Endocrine System Diseases
MeSH Terms: conditions — Endocrine System Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
AIMS AND OBJECTIVES

1. To evaluate whether acute pancreatitis results in increased endocrine dysfunction or not?
2. To evaluate whether severity of acute pancreatitis have an impact on the development of endocrine dysfunction or not?

1.4 MATERIALS AND METHODS:- Definitions … 1) Acute pancreatitis…..Acute pancreatitis is best defined clinically by a patient presenting with 2 of the following 3 criteria: (1) symptoms(e.g., epigastric pain) consistent with pancreatitis, (2) a serum amylase or lipase level greater than 3 times the laboratory's upper limit of normal, and (3) radiologic imaging consistent with pancreatitis, usually using CT or MRI.The AtlantaCriteria revision of 2012 classifies severity as mild, moderately severe, or severe. Mild acute pancreatitis has no organ failure, no local or systemic complications.Moderately-severe acute pancreatitis is defined by the presence of transient organ failure (lasting <48 hours) and/or local complications.Severe acute pancreatitis is defined by persistent organ failure (lasting >48 hours). Local complications include peripancreatic fluid collections, pancreatic and peripancreatic necrosis (sterile or infected), pseudocyst, and walled-offnecrosis (sterile or infected) .

Prediabetes/Diabetes….Prediabetes is defined by fasting blood glucose (FBG ≥(100 mg/dL) and <(126 mg/dL),and/or 2 h oral glucose tolerance test (OGTT) criteria as >/ (140 mg/dL) and < (200 mg/dL)) or HbA1c of 5.7% to 6.4%. DM is defined as (FBG ≥ (126 mg/dL) or 2 hOGTT ≥ (200 mg/dL)or HbA1c value>/ 6.5% ,treatment with insulin, oral hypoglycaemic agents or specific dietary management. Diagnosis of diabetes in asymptomatic patients is established by presence of abnormal test results in 2 out of 3 parameters used(FBG,OGTT or HbA1c) or if only one test result is abnormal ,needs to be confirmed on next day or few days later by repeat testing of the specific parameter.

Study design :- Single center ,prospective cohort study performed at a tertiary care centre (Asian institute of gastroenterology , Hyderabad) from Feb 2019 to May 2020.

Participant recruitment procedures…. Patient enrollment from Feb 2019 to May 2019 & follow up of each case upto 1 year, upto May 2020(1 year follow up).

Primary outcome-Development of endocrine dysfunction (diabetes & prediabetes) after acute pancreatitis Secondary outcomes-Whether severity of acute pancreatitis correlate with development of diabetes & prediabetes.

DETAILED DESCRIPTION:
METHODOLOGY: Patients of acute pancreatitis will be screened as per inclusion/exclusion criteria and patients with first episode of acute pancreatitis who meet the ATLANTA definition, will be graded for severity as per Modified Marshall criteria. Control group for the study will include nondiabetic /non prediabetic volunteers who come to OPD for master health check up or who are being suspected to have functional syndromes like functional dyspepsia or irritable bowel syndrome.The study will be a prospective cohort study in which initial recruitment will be for 4 months from Feb 2019 to May 2019, & recruited patients will be followed for a period of 1 year each from the period of recruitment, and as such the study is expected to complete by May 2020. On admission in addition to routine blood investigations , specific investigations for acute pancreatitis will be done(complete details in proforma) which include serum amylase ,serum lipase, USG abdomen, CECT abdomen(after 72hrs of onset of acute pancreatitis) will be done to assess for pancreatic necrosis. Blood sugar (fasting, postprandial) & HBA1c will be done on admission to evaluate the diabetic status of the patient. C peptide and Fasting insulin levels which will help assess the insulin resistance will be done at onset only in these patients .Control group will be assessed clinically and only clinically relevant investigations in addition to blood sugar (fasting, postprandial) & HBA1c will be done at initiation & at 6months & 1 year of follow up(follow up will be via telephonic communication or if possible in person) On follow up at 2months , 6months & 12 months patients will be reassessed either in person (if possible) or via telephonic communication for endocrine dysfunction , which will be assessed by simple and routine tests as mentioned ( Blood sugar-fasting, postprandial & HbA1c).Controls will be clinically assessed and if clinically stable and asymptomatic will be assessed for diabetic status only with Blood sugar (fasting, postprandial) & HBA1c at initiation & subsequently at 6 months and 1 year end.

Statistical analysis :Data will be collected using a structured study proforma. Data will be put in MS EXCEL for further analysis .Results will be expressed as mean(SD), median (IQR) for continuous variables and percentage for categorical variables etc. Appropriate parametric and non parametric will be applied. SPSS (21st version) will be used for statistical analyses.

Primary outcome…. To estimate incidence of endocrinopathy (diabetes & prediabetes)among Acute Pancreatitis patients.

ELIGIBILITY:
Inclusion Criteria:

1 )Ist episode of acute pancreatitis. 2) Non diabetic or non pre diabetic as per American Diabetes Association criteria .

3) Age >18yrs.

Exclusion Criteria:

1. Acute pancreatitis cases who die within 1 month of hospitalization.
2. Recurrent acute pancreatitis
3. Chronic pancreatitis.
4. Previous diagnosed diabetes or prediabetes
5. Any malignancy
6. Age <18yrs
7. Pregnant females or lactating women.
8. Chronic diarrhea, intestinal tuberculosis or Crohns disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Required sample size is 90 subjects with 80% power and 0.05 as type 1 error.
Sampling Method: Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-05-31 (Actual); Study Completion 2020-08-30 (Estimated)

PRIMARY OUTCOMES:
Development of endocrine dysfunction (diabetes & prediabetes) after acute pancreatitis | 1 year
  Prediabetes/Diabetes is defined by fasting blood glucose (FBG ≥(100 mg/dL),HbA1c value>/ 6.5% ,

SECONDARY OUTCOMES:
2) To evaluate whether severity of acute pancreatitis have an impact on the development of endocrine dysfunction or not? | 72 hours
  Severity of acute pancreatitis can be done based on elevated serum amylase and lipase levels.normal range of amylase level is( 28-100 units U/I) more than 3 times of normal range indicated acute pancreatitis, normal range of lipase is (5.6-51.3) more than 3 times of normal range leads to acute pancreatitis.

CONTACTS AND LOCATIONS:
Overall Officials: Dr MANU TANDAN, MBBS MD DM, Principal Investigator — Asian Institute of Gastroenterology, India
Locations (1):
- Asian Institute of Gastroenterology/AIG Hospitals, Hyderabad, Telangana, India